# Intervention for Battered Sheltered Women With Substance Use Randomized Trial

NCT02629133

March 15, 2017

#### **Statistical Analyses**

### **Statistical Analysis Overview**

- 1. Descriptively characterize the: (a) **feasibility** of the SHE Program, and the (b) **acceptability** via participant report of ease of use, helpfulness, and overall satisfaction.
- 2. Examine preliminary evidence that relative to control condition, the computer-based intervention (SHE) will result in improvements in our primary outcomes of substance use (heavy drinking or drug using) days over a 6-month postshelter period and in our secondary outcomes of greater use of substance use services (both treatment and self-help utilization) and reduced IPV severity over a 6-month postshelter period. Theorized mediators include readiness to change and self-efficacy for behaviors related to substance use.

#### **Comparison Group Selection**

SHE intervention Control condition

#### Comments

Assessment of feasibility and acceptability of the intervention and research procedures is the project's primary goal. However, pilot data can be used to demonstrate whether the effects of treatment look promising across a set of outcome variables. We will obtain the between treatment condition effect size estimates at each assessment and the correlation between the same dependent variable at adjacent assessments. A sample of ~20-21 in each condition should provide some information relevant to demonstrating potential promise for the intervention.

#### Type of Statistical Test [\*]

Other (primary analyses focus on feasibility and acceptability)

#### Comments [\*]

Secondary analyses will explore differences between conditions on outcome variables.

**Statistical Test of Hypothesis** (or Method of Estimation or Other Statistical Analysis required) We will calculate the effect sizes and 95% confidence intervals for intervention effects on outcomes using hierarchical linear modeling with a tightly constrained covariance structure. However, this is not primarily a hypothesis-testing study.

#### P-Value [\*]

There is no null hypothesis. If we use any p-value, it will be .05.

#### Comments

None

#### Method [\*]

We will calculate the effect sizes and 95% confidence intervals for intervention effects on outcomes using hierarchical linear modeling with a tightly constrained covariance structure.

Baseline values of each outcome variable will serve as a covariate in analyses. However, primary results are descriptive results of feasibility and acceptability.

## Other Method Name [\*] None **Comments** None Method of Estimation (or Statistical Test of Hypothesis or Other Statistical Analysis required) NA **Estimation Parameter** [\*] Other Parameter Name [\*] Estimated Value [\*] NA **Confidence Interval** (*If applicable*) 95% Level [\*] NA Number of Sides [\*] 2-sided. Lower Limit [\*] NA Upper Limit [\*] NA NA (Not Available) Explanation [\*] This is not relevant to our analysis **Parameter Dispersion Type**

Standard Error of the Mean

## **Dispersion Value**

Standard Deviation

NA

#### **Estimation Comments**

NA

## **Other Statistical Analysis**

NA